CLINICAL TRIAL: NCT05036057
Title: Investigation of the Psychometric Properties of the Turkish Version of the Individual Knowledge Statement Questionnaire of Chronic Obstructive Pulmonary Disease (COPD) Patient and Resident Proxies
Brief Title: Turkish Version of the Individual Knowledge Statement Questionnaire of Chronic Obstructive Pulmonary Disease (COPD)
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Izmir Katip Celebi University (Other)
Collaborators: Izmir Dr Suat Seren Chest Diseases and Surgery Education and Research Hospital (Other)
Responsible Party: Principal Investigator, Ilknur Naz, Associate Professor, Izmir Katip Celebi University
Other Study IDs: 2021-GOKAE-0221
Record Dates: First submitted 2021-09-02; First posted 2021-09-05 (Actual); Last update posted 2021-09-05 (Actual); Status verified 2021-09

CONDITIONS: Chronic Obstructive Pulmonary Disease; Knowledge, Attitudes, Practice
Keywords: COPD; patient knowledge; proxies
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Behavior | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 15 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- COPD patients and their proxies: Patients will do the Individual Knowledge Statement Questionnaire of Chronic Obstructive Pulmonary Disease (COPD), the COPD Assesment Test (CAT), the Saint George Respiratory Disease Questionnaire (SGRQ), the Charlson Comorbidity Index, and will rate the disease and general knowledge level on a numerical scale.
  Proxies of patients will do the Individual Knowledge Statement Questionnaire of Chronic Obstructive Pulmonary Disease (COPD) and will rate the disease and general knowledge level on a numerical scale.
  Interventions: Other: Questionnaire

INTERVENTIONS:
Other: Questionnaire — Patients will do the Individual Knowledge Statement Questionnaire of Chronic Obstructive Pulmonary Disease (COPD), the COPD Assesment Test (CAT), the Saint George Respiratory Disease Questionnaire (SGRQ), the Charlson Comorbidity Index, and will rate the disease and general knowledge level on a numerical scale.
  Proxies of patients will do the Individual Knowledge Statement Questionnaire of Chronic Obstructive Pulmonary Disease (COPD) and will rate the disease and general knowledge level on a numerical scale.

SUMMARY:
The Individual Knowledge Statement Questionnaire of Chronic Obstructive Pulmonary Disease (COPD) Patient and Resident Proxies questionnaire, which can be used in patients with Chronic Obstructive Pulmonary Disease (COPD) and their relatives, will be adapted into Turkish and its psychometric properties will be examined, and the knowledge level of patients and their relatives about the disease and general health will be investigated.

DETAILED DESCRIPTION:
The socio-demographic characteristics of the patients and their relatives will be obtained by asking to them by mutual interview method.

A disease-specific test, the COPD Assessment Test (CAT), will be used to assess patients' own health, and the St George Respiratory Questionnaire (SGRQ) will be used to assess patients' quality of life.

Comorbidities reported by the patient and their relatives will be filled in the Charlson Comorbidity Index. The dyspnea that patients encounter in their daily lives will be questioned with the Modified Medical Research Council (mMRC) Dyspnea Scale.

The "Individual Knowledge Statements of Patients and Resident Proxies" will be used for the individual information of the patient and their relatives about the disease and general health.

There is no control group in the study. SGRQ, CAT and numerical rating scale will be used for the validity of the Turkish version of Individual Knowledge Statements of Patients and Resident Proxies. For the test-retest, the evaluation will be done again after 15 days.

ELIGIBILITY:
Inclusion Criteria:

* Being 18 years or older
* Being diagnosed with COPD by a specialist physician (for patients)
* Being clinically stable (For patients, no history of hospital admission/hospitalization due to exacerbation in the last 4 weeks)
* Having information about the diagnosis (For patients)
* To read, write and understand Turkish
* Volunteering to participate in the study
* Being a proxy of the patient (living with the patient regardless of whether they are providing care or not)

Exclusion Criteria:

* Having musculoskeletal, neurological, cardiac, and/or cognitive problems other than COPD, which may create a caregiver burden for the patient's relative

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Study population will be patient with diagnosed COPD in the Chest Diseases Outpatient Clinic of Dr Suat Seren Chest Diseases and Surgery Training and Research Hospital, and their proxies.
Sampling Method: Probability Sample
Enrollment: 340 (Estimated)
Dates: Start 2021-10-04 (Estimated); Primary Completion 2021-11-25 (Estimated); Study Completion 2022-10-04 (Estimated)

PRIMARY OUTCOMES:
Individual Knowledge Statement Questionnaire of Chronic Obstructive Pulmonary Disease (COPD) | Baseline
  The scale is a 34-item questionnaire that evaluates the knowledge of COPD patients and their relatives about the disease and general health.
  All of 34 statements can be answered as "true", "false" or "don't know". A score out of 34 points will be obtained by giving 1 point to each correct answer appropriate to the question.
  Higher score will show more knowledge level. It will done by patients and their proxies.

SECONDARY OUTCOMES:
COPD Assesment Test (CAT) | Baseline
  The COPD Assessment Test (CAT) is a questionnaire, which consist of 8 questions, for people with COPD. It is designed to measure the impact of COPD on a person's life, and how this changes over time. The eight questions are each rated on a scale of 0 to 5. Range of CAT scores from 0-40. Higher scores denote a more severe impact of COPD on a patient's life. It will done by patients.
The modified Medical Research Council (mMRC) scale | Baseline
  The mMRC scale is a self-rating tool to measure the degree of disability that breathlessness poses on day-to-day activities on a scale from 0 to 4: 0, no breathlessness except on strenuous exercise; 1, shortness of breath when hurrying on the level or walking up a slight hill; 2, walks slower than people of same age on the level because of breathlessness or has to stop to catch breath when walking at their own pace on the level; 3, stops for breath after walking ∼100 m or after few minutes on the level; and 4, too breathless to leave the house, or breathless when dressing or undressing.
  It will done by patients.
Charlson Comorbidity Index | Baseline
  The Charlson Comorbidity Index is a method of categorizing comorbidities of patients based on the International Classification of Diseases (ICD) diagnosis codes found in administrative data, such as hospital abstracts data. Each comorbidity category has an associated weight (from 1 to 6), based on the adjusted risk of mortality or resource use, and the sum of all the weights results in a single comorbidity score for a patient. A score of zero indicates that no comorbidities were found. The higher the score, the more likely the predicted outcome will result in mortality or higher resource use.
The St George's Respiratory Questionnaire (SGRQ) | Baseline
  The St George's Respiratory Questionnaire (SGRQ) is a validated, commonly used questionnaire for measuring quality of life in patients with chronic obstructive pulmonary disease (COPD). It consists of 76 items in three domains (symptoms, activity, impact of disease on daily life).
  A total score of SGRQ is calculated from 0 (no health impairment) to 100 (maximum health impairment). There are also the score of each domain are scored from 0 to 100.
Knowledge Score 0-10 Numerical Rating | Baseline
  The 11-point numeric scale ranges from '0' (e.g. "nothing known") to '10' (e.g. "maximal knowledge").
  It can be administered verbally. Scores range from 0-10 points, with higher scores indicating greater knowledge. It will done by patients and their proxies. They will be asked to rate their level of knowledge about COPD and general health.
The Sociodemographic Characteristics | Baseline
  The sociodemographic characteristics of the patient and their relatives will be recorded in the registration form.
  Socio-demographic information will be asked from people and their relatives by mutual interview method.
  Age, gender, marital status, education level, occupation, medical history, duration of COPD, regularly used medications - oxygen support - non-invasive mechanical ventilation (NIMV), smoking status, alcohol consumption, exercise habits, attacks and pulmonary rehabilitation histories will be questioned in this section.